CLINICAL TRIAL: NCT01473316
Title: An Open-Label, Fixed-Sequence, 2-Period Study to Determine the Effect of Ketoconazole on the Pharmacokinetics of GDC-0980
Brief Title: Study to Determine the Effect of Ketoconazole on the Pharmacokinetics of GDC-0980
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP27913
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one; Ketoconazole

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0980; Drug: Ketoconazole

INTERVENTIONS:
Drug: GDC-0980 — Single oral dose
Drug: Ketoconazole — Repeating Oral Dose

SUMMARY:
This will be an open-label, fixed-sequence, single-center, 2 period study. The study is designed to determine the effect of ketoconazole on the pharmacokinetics of GDC-0980.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal and/or surgically sterile adult nonsmoking female subject between 18 and 65 years of age, inclusive, with a body mass index of 18 to 32 kg/m2, inclusive
* Medically healthy as determined by the absence of clinically significant findings in the physical examination, medical history, vital sign measurements, clinical laboratory tests, or 12 lead electrocardiograms (ECGs) as determined by the investigator
* Female subject of nonchildbearing potential

Exclusion Criteria:

* History or clinical manifestations of significant metabolic (including type 1 and 2 diabetes), hepatic, renal, hematological (including hypercholesterolemia and triglyceridemia), pulmonary, cardiovascular, endocrine, gastrointestinal (including gastric or duodenal ulcers), urological, neurological, or psychiatric disorders, or cancer
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of severe physical injury, direct impact trauma, or neurological trauma within 6 months before Day 1 of Period 1
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of stomach or intestinal surgery or resection that could potentially alter absorption and/or excretion of orally administered drugs, with the exception of appendectomy, hernia repair, and cholecystectomy, which are allowed
* History of active liver disease, including hepatitis or cirrhosis
* History or presence of an abnormal ECG
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* Abnormality on the chest x-ray at Screening determined to be clinically significant by the investigator and medical monitor
* History of alcoholism, drug abuse, or drug addiction
* Used any nicotine-containing or nicotine-replacement products within 6 months before Day 1 of Period 1
* Participated in any other investigational drug study in which receipt of an investigational study drug occurred within 1 month or 5 half-lives before Day 1 of Period 1
* Used any prescription medications/products including monoamine oxidase inhibitors, thioridazine, pimozide, or antidepressants within 1 month (2 weeks for antibiotics) before Day 1 of Period 1, with the exception of hormone replacement therapy or 2 weeks' use of narcotics for pain, unless deemed acceptable by the investigator
* Used medications capable of inhibiting hepatic enzymes within 1 month or 5 half-lives before Day 1 of Period 1
* Received any vaccination or immunization within 1 month before Day 1 of Period 1
* Used proton pump inhibitors or histamine H2 receptor antagonists within 1 month before Day 1 of Period 1
* Known hypersensitivity to ketoconazole, or other azole antifungals
* Used any over-the-counter, nonprescription preparations within 7 days before Day 1 of Period 1, unless deemed acceptable by the investigator
* Used alcohol-containing, grapefruit-containing, or caffeine containing foods or beverages within 72 hours before Day 1 of Period 1, unless deemed acceptable by the investigator
* Poor peripheral venous access
* Donated blood within 2 weeks or plasma within 1 week before Day 1 of Period 1
* Received blood products within 2 months before Day 1 of Period 1
* Positive urine drug or alcohol screen
* Positive screen for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus types 1 and 2
* Diagnosed with a vitamin B12 deficiency
* Any acute or chronic condition that, in the opinion of the investigator, would limit the subject's ability to complete or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: maximum observed plasma concentration | Up to approximately 10 days
Pharmacokinetics: time to reach maximum observed plasma concentration | Up to approximately 10 days

SECONDARY OUTCOMES:
Adverse events | Up to approximately 40 days
Clinical laboratory test results (hematology and serum chemistry) | Up to approximately 10 days
Vital sign measurements (sitting systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature) | Up to approximately 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Austin, Texas, United States